CLINICAL TRIAL: NCT00349206
Title: Phase 1 Study of the Combination of BAY 43-9006 (Sorafenib) and CCI-779 (Temsirolimus) in Patients With Metastatic Melanoma
Brief Title: Sorafenib and Temsirolimus in Treating Patients With Metastatic, Recurrent, or Unresectable Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00131; NCI-2009-00131 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2005-0215; CDR0000480157; 2005-0215 (Other: M D Anderson Cancer Center); 7149 (Other: CTEP); P30CA016672 (NIH); N01CM62202 (NIH)
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2013-02

CONDITIONS: Melanoma; Recurrent Melanoma; Stage III Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Sorafenib; temsirolimus; Sirolimus

ARMS (1):
- Arm 1 (Experimental): Patients receive temsirolimus IV over 30 minutes on days 1, 8,15, and 22 and oral sorafenib once or twice daily on days 1-28.
  Interventions: Drug: sorafenib tosylate; Drug: temsirolimus

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel

SUMMARY:
This phase I trial is studying the side effects and best dose of temsirolimus when given together with sorafenib and to see how well they work in treating patients with metastatic, recurrent, or unresectable melanoma. Sorafenib and temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sorafenib may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving sorafenib together with temosirolimus may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of temsirolimus when administered with sorafenib in patients with metastatic, recurrent, or unresectable melanoma.

II. To determine the safety and toxicity of this regimen in these patients.

SECONDARY OBJECTIVES:

I. To Determine the population pharmacokinetics of this regimen in these patients.

II. To correlate tumor and blood biomarkers with clinical outcome in patients treated with this regimen.

OUTLINE: This is a multicenter, phase I, dose-escalation study followed by a phase II, open-label study (2005-0215).

Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22 and oral sorafenib once or twice daily on days 1-28. Treatment course repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3-6 months.

ELIGIBILITY:
Criteria:

* Histologically or cytologically confirmed melanoma, meeting 1 of the following criteria: recurrent or unresectable stage III disease, stage IV disease, non-choroidal origin.
* Tumor must be accessible to biopsy unless appropriate tumor sample collection has occurred within the past 3 months and patient agrees to provide these samples for this study.
* ECOG performance status 0-1.
* Bilirubin normal
* Creatinine normal or creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after completion of study treatment.
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to sorafenib or temsirolimus.
* No uncontrolled hypertension, defined as systolic blood pressure > 140 mm Hg on 2 separate days < 1 week prior to study entry OR diastolic pressure > 90 mm Hg on 2 separate days < 1 week prior to study entry.
* No evidence of bleeding diathesis or coagulopathy.
* No condition that would impair the ability to swallow pills (e.g., gastrointestinal tract disease resulting in an inability to take oral medication; requirement for IV alimentation; or active peptic ulcer disease).
* No uncontrolled illness including, but not limited to, any of the following: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness or social situations that would limit study compliance.
* No traumatic injury within the past 3 weeks.
* No more than 1 prior systemic chemotherapy regimen for metastatic melanoma (Phase II).
* No prior sorafenib, temsirolimus, or any other agents targeting raf, vascular endothelial growth factor (VEGF)/VEGF receptor, or mTOR (Phase II).
* No prior surgical procedures affecting absorption.
* At least 3 weeks since prior major surgery.
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) for melanoma and recovered.
* At least 4 weeks since prior radiotherapy and recovered.
* Prior biologic or immunotherapeutic regimens allowed.
* Prior regional chemotherapy regimens (e.g., isolated limb perfusion) allowed but only 1 prior regional chemotherapy regimen allowed if all target lesions are within the prior regional treatment field.
* No concurrent enzyme-inducing antiepileptic drugs including, but not limited to, any of the following: phenytoin, carbamazepine, phenobarbital, rifampin or Hypericum perforatum (St. John's wort).
* No concurrent prophylactic hematopoietic colony-stimulating factors.
* No other concurrent investigational agents.
* No other concurrent anticancer agents or therapies for this cancer.
* No concurrent full-dose anticoagulation (i.e., warfarin, IV heparin, or low-molecular weight heparin).
* No concurrent grapefruit or grapefruit juice.
* No concurrent combination antiretroviral therapy for HIV-positive patients.
* Concurrent prophylactic anticoagulation therapy (e.g., low-dose warfarin) allowed provided PT INR < 1.1 times ULN.
* Unidimensionally measurable disease >= 20 mm by conventional techniques or >= 10 mm by spiral CT scan (longest diameter to be recorded) and margins of visible cutaneous metastatic lesions should be clearly defined and measured in at least one dimension as >= 10 mm.
* No known brain metastases unless the following criteria are met: no radiographical evidence of recurrences in the brain >= 3 months after complete resection of the brain metastases, asymptomatic brain metastases stable for >= 3 months since whole-brain radiation therapy and/or stereotactic radiosurgery and must not require steroid for brain metastases.
* WBC >= 3,000/mm³
* Absolute neutrophil count >= 1,500/mm³
* Platelet count >= 100,000/mm³
* Serum cholesterol =< 350 mg/dL
* Triglycerides =< 400 mg/dL
* AST/ALT =< 2.5 times upper limit of normal.
* No peripheral neuropathy > grade 2.
* At least 5 years since prior chemotherapy for other types of cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2006-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of CCI-779 in combination with BAY43-9006 (Phase I) determined by DLT assessed by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase I) | 28 days
Objective response rate (complete response and partial response) CCI-779 in combination with BAY43-9006 (Phase II) | Up to 5 years

SECONDARY OUTCOMES:
Progression-free survival | The duration of time from start of treatment to date of first evidence of progression or the date of last follow-up for patients who do not progress, assessed up to 5 years
  Kaplan-Meier life table methods and Cox proportional hazards regression modeling will be utilized to analyze progression-free survival and overall survival.
Overall survival | 5 years
  Kaplan-Meier life table methods and Cox proportional hazards regression modeling will be utilized to analyze progression-free survival and overall survival.
Noncompartmental pharmacokinetic parameters of BAY43-9006 and CCI-779 estimated using a validated commercial software | Week 1 and 3
  Maximum concentration (Cmax) and time to Cmax (tmax) will be the observed values. Area under the plasma concentration-time curve from zero to last observable time (AUClast).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kim, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States